CLINICAL TRIAL: NCT01025869
Title: The Clinical Evaluation of the Cinatra™ Corolimus-Eluting Coronary Stent in De Novo Lesions in Native Coronary Arteries
Acronym: VANTAGE-1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated following completion of 2 year time point: Sponsor decision
Sponsor: Atrium Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 902
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stent System (Other): Cinatra™ Corolimus Eluting Coronary Stent System
  Interventions: Device: Cinatra™ Corolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: Cinatra™ Corolimus Eluting Coronary Stent System — Stent implantation

SUMMARY:
To investigate the safety and efficacy of the Cinatra™ Corolimus Drug Eluting Stent for the treatment of de novo lesions in native coronary arteries.

DETAILED DESCRIPTION:
This is a single-arm, multicentre pilot study designed to provide an indication of the effectiveness and safety of the Cinatra™ Corolimus Eluting Coronary Stent System. The primary endpoint to be evaluated in this study is late lumen loss (in-stent) at 6 months post-procedure as measured by QCA in the 30 participants undergoing angiography at this timepoint. Late lumen loss is defined as the difference between the post-index procedure minimal lumen diameter (MLD) and the follow-up MLD.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years old
2. Patient is an acceptable candidate for percutaneous coronary intervention (PCI), stenting, and emergent coronary artery bypass graft (CABG) surgery
3. Patient has clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia, and/or a positive functional study
4. Female subjects of childbearing potential must have a negative pregnancy test within 7 days before the trial procedure
5. Patient or subject's legal representative has been informed of the nature of the trial and agrees to its provisions and has provided written informed consent as approved by the Hospital Research Ethics Committee (HREC) of the respective investigational site
6. Patient agrees to comply with specified follow-up evaluations and to return to the same investigational site where the procedure was performed

Angiographic:

1. Patient has either a single target lesion, or two lesions (target and non-target) located in separate coronary arteries
2. If a non-target lesion is treated, it must be treated first and only with commercially available PTCA balloons and/or stents. Post PCI of the non-target vessel, all of the following conditions must be met:

   * Residual diameter stenosis <10%
   * Absence of any angiographic complications
   * Absence of ischaemic symptoms
   * Absence of significant new arrhythmia or ECG monitoring changes suggestive of ischaemia
3. Target lesion must be a de novo lesion in native coronary artery
4. Target lesion must be ≤ 22 mm in length
5. Target lesion must have a stenosis of ≥ 50% and < 100%
6. Target vessel must have a reference vessel diameter (RVD) appropriate for treatment with a of 3.0mm or3.5 mm stent
7. Target vessel must have a Thrombolysis in Myocardial Infarction (TIMI) flow ≥ 2

Exclusion Criteria:

1. Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, cobalt, chromium, stent coatings (i.e. fatty acids, glycerides, and alpha tocopherol), or a sensitivity to contrast media, which cannot be adequately pre-medicated
2. History of an allergic reaction or significant sensitivity to drugs such as , zotarolimus, rapamycin, tacrolimus, everolimus, or any other analogue or derivative
3. Platelet count < 100,000 cells/mm³ or > 700,000 cells/mm³, or a white blood cell (WBC) count < 3,000 cells/mm³ within 7 days prior to index procedure
4. Serum creatinine level 170 micromol/L within 7 days prior to index procedure
5. Evidence of an acute myocardial infarction (MI) within 72 hours of the intended trial procedure (defined as: Q wave myocardial infarction (QWMI) or non-Q wave myocardial infarction (NQWMI) having CK enzymes > 2X the laboratory upper limit of normal with the presence of an elevated CK-MB (any amount above the laboratory upper limit of normal)
6. Previous PCI of the target vessel within 9 months prior to the procedure
7. Any planned additional PCI procedure within 30 days post-index procedure and/or planned PCI of the target vessel within 12 months post-procedure
8. During the index procedure, the target and/or non-target lesion(s) requires treatment with a device other than PTCA prior to stent placement (including, but not limited to, cutting balloon, atherectomy, thrombectomy, etc.)
9. Left ventricular ejection fraction (LVEF) < 30% if evaluated, or clinical evidence of significant congestive heart failure (NYHA Class III or IV) within the prior 30 days
10. History of a stroke or transient ischemic attack (TIA) within the prior 6 months
11. Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months
12. History of bleeding diathesis or coagulopathy or will refuse blood transfusions
13. Concurrent medical condition with a life expectancy of less than 12 months
14. Any previous treatment of the target vessel(s) for restenosis, including brachytherapy

16. Any condition which, in the Investigator's opinion, may interfere with the subject's optimal participation in the study 17. Currently participating in an investigational drug or another device trial that has not completed the primary endpoint or that clinically interferes with the current trial endpoints; or requires coronary angiography, IVUS or other coronary artery imaging procedures

Angiographic:

1. Target lesion is located in native vessel distal to anastomosis with a saphenous vein graft or a left/right internal mammary artery (LIMA/RIMA) bypass with more than 40% diameter stenosis anywhere within the graft
2. Previous stenting in the target vessel.
3. The target vessel has other lesions with greater than 40% diameter stenosis based on visual estimate or on-line QCA
4. The target vessel has evidence of thrombus
5. The target vessel is excessively tortuous (two bends > 90º to reach the target lesion)
6. The target lesion has any of the following characteristics:

   * Lesion location is aorto-ostial, an unprotected left main lesion, or within 5 mm of the origin of the left anterior descending (LAD) or left circumflex (LCX)
   * Involves a side branch > 2.0 mm in diameter
   * Is at or distal to a > 45º bend in the vessel
   * Is severely calcified
7. Unprotected left main coronary artery disease (an obstruction greater than 50% in the left main coronary artery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-12; Primary Completion 2010-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
In-stent late lumen loss (LLL) as measured by quantitative coronary angiography (QCA). | 6 months post treatment

SECONDARY OUTCOMES:
Target lesion revascularization | 1, 6 and 18 month and annually to 5 years
Target vessel revascularization | 1 month and at all follow up to 5 years
Stent thrombosis | All follow ups
Neointimal Hyperplasia | 6 and 18 months
Binary restenosis | 6 and 18 months
MACE (Major Adverse Cardiac Event) | 1 month, 6 month, 18 month and annually to 5 years
In-segment late lumen loss (LLL) as measured by quantitative coronary angiography | 6 and 18 months
In-stent late lumen loss (LLL) as measured by quantitative coronary angiography | 18 months (optional)
Minimal Lumen Diameter (MLD), in-stent and in-segment | 6 and 18 months
Rates of incomplete stent apposition | 6 and 18 months
Device success defined as achievement of a final residual diameter stenosis of < 30% measured by QCA, using the study device only. | procedure
Lesion treatment success is defined as <30% residual stenosis measured by QCA by any treatment | Procedure
Procedure success defined as lesion success without the occurrence of MACE during the hospital stay | discharge

CONTACTS AND LOCATIONS:
Overall Officials: John Ormiston, MD, Principal Investigator — Associate Professor and Interventional Cardiologist at Auckland City Hospital
Locations (4):
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Mercy Angiography, Auckland
  - North Shore Hospital, Auckland
  - Christchurch Hospital, Christchurch